CLINICAL TRIAL: NCT07136220
Title: A Pilot Study to Evaluate Equol and Its Effects on Menopausal Symptoms Experienced by Women in Singapore
Acronym: EQUOL
Status: Recruiting | Type: Observational
Sponsor: Ang Seng Bin (Other Government)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Ang Seng Bin, Senior Consultant, KK Women's and Children's Hospital
Organization: KK Women's and Children's Hospital (Other Government)
Other Study IDs: 2025/0693
Record Dates: First submitted 2025-08-08; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Menopause
Keywords: menopause; equol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Consumption of soy protein bar — The participants will be provided one soy protein bar to consume after dinner on day 1.

SUMMARY:
The main aim of this study is to evaluate the effect of equol on menopausal symptoms of women. Our hypothesis is that equol producers will have milder menopausal symptoms compared to non-equol producers. Equol is known as a metabolite produced by gut microbiota from soy-related diet and has estrogen-like activity compared to the isoflavones from soybean.

Previous studies have shown that some women can produce equol from soy-related diet, but the others cannot because they don't have the bacteria which can metabolite daidzein in gut even if they take isoflavones thorough soybean products.

This study will involve participants consuming a soy protein bar and collection of urine samples before and after its consumption.

DETAILED DESCRIPTION:
Day 0 - Recruitment and consent taking. Height, weight and blood pressure would be measured. Patients will also fill up questionnaires on basic demographics, menopausal symptoms (Menopause Rating Scale and Vulvovaginal Symptom Questionnaire), Food Frequency Questionnaire for Soy intake, International Physical Activity Questionnaire.

Day 1 - Collect first morning urine between 5ml to 10 ml in the pre-labelled (will not contain identifiers but only assigned study subject number) containers provided. Store the urine sample in cool place in room temperature and dispatch to site after the second sample has been collected. To consume a soy based protein bar provided by study after dinner on day 1.

Day 2 - Collect first morning urine between 5ml to 10 ml in the pre-labelled(will not contain identifiers but only assigned study subject number) containers provided. Double bag the containers and call courier to dispatch urine to KK Women's and Children's Hospital.

All urine samples received will be immediately frozen and stored in KKH in a freezer. The samples will be couriered to Saga Nutraceuticals Research Institute, Otsuka Pharmaceutical Co. Ltd, Japan in batches for analysis of urinary equol concentration. Clinical Trials Agreement has been executed between Otsuka Pharmaceutical Co. Ltd, Japan and KK Women's and Children's Hospital.

ELIGIBILITY:
Inclusion Criteria:

- Women aged 40-60

Exclusion Criteria:

* Pregnant women
* Allergy to Soy
* Allergy to nuts
* Consumed antibiotics within 7 days of the study
* Has a history of autoimmune diseases
* Has a history of thyroid disease
* On medical treatment with hormone therapy, elective oestrogen receptors modulators
* Consuming equol-containing supplements or food
* Consuming painkillers
* Consuming anti-depressants and/or sleeping pills

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women in Singapore aged 40-60
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Urine Equol Concentration | first morning urine sample collected at baseline and first urine sample collected the morning after consuming the soy bar
  Equol is a metabolite of isoflavone which is secreted in the urine

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu B, Qin L, Liu A, Uchiyama S, Ueno T, Li X, Wang P. Prevalence of the equol-producer phenotype and its relationship with dietary isoflavone and serum lipids in healthy Chinese adults. J Epidemiol. 2010;20(5):377-84. doi: 10.2188/jea.je20090185. Epub 2010 Jul 24. PMID 20671375
- [Background] Tseng M, Byrne C, Kurzer MS, Fang CY. Equol-producing status, isoflavone intake, and breast density in a sample of U.S. Chinese women. Cancer Epidemiol Biomarkers Prev. 2013 Nov;22(11):1975-83. doi: 10.1158/1055-9965.EPI-13-0593. Epub 2013 Sep 9. PMID 24019393

DOCUMENTS (1):
  • Informed Consent Form (2025-06-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT07136220/ICF_000.pdf